CLINICAL TRIAL: NCT04686318
Title: What is the Diagnostic and Prognostic Accuracy of C-reactive Protein, Serum Procalcitonin and Soluble Urokinase Plasminogen Activator Receptor in the Initial Investigation of Patients With Suspected Acute Pyelonephritis
Brief Title: Accuracy of Infection Biomarkers in the Investigation of Patients With Suspected Acute Pyelonephritis
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-12c-2020
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Acute Pyelonephritis
Keywords: C-reactive protein; serum procalcitonin; soluble urokinase plasminogen activator receptor; diagnostic and prognostic markers; emergency department
MeSH Terms: conditions — Disease; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspected acute pyelonephritis: All patients admitted to the emergency department with suspected acute pyelonephritis assessed by the receiving physician
  Interventions: Diagnostic Test: Biomarkers for acute pyelonephritis

INTERVENTIONS:
Diagnostic Test: Biomarkers for acute pyelonephritis — Blood samples will be collected by a medical laboratory technologist and transferred to the local laboratory for analysis of CRP, PCT and suPAR. Laboratory staff will be blinded to participant diagnosis and outcome. CRP and PCT results will be available to the treating physician, but the suPAR result will not be available.
  * Diagnostic test of CRP. CRP will be measured using an immunoturbidimetric assay (Tina-quant®, Roche) on Roche/Hitachi Cobas© systems.
  * Diagnostic test of PCT: Plasma PCT will be quantified by an automated sandwich immunoassay "ECLIA" (Elecsys®, BRAHMS PCT-analyses) on Cobas© within two hours from collection according to standard procedure.
  * Diagnostic test of suPAR: Plasma suPAR will be quantified by using the commercial available suPARnostic© Tubilatex assay reagents (ViroGates, Denmark) on Cobas© as previously validated (35). Separated plasma is kept refrigerated and analysed for suPAR within 48 hours after collection.

SUMMARY:
The aim of this study is to investigate the diagnostic and prognostic value of C-reactive protein (CRP), serum procalcitonin (PCT) and soluble urokinase plasminogen activator receptor (suPAR) in the initial investigation of patients hospitalized with suspected acute pyelonephritis (APN).

DETAILED DESCRIPTION:
Acute pyelonephritis (APN) is a severe acute infection in the upper urinary tract, which quite frequently is seen in the emergency department (ED). In our study, we define APN as a urinary tract infection with extension above the bladder, implicated by systemic affection in a suspected urinary tract infection (ie, fever, chills, malaise and/or lethargy beyond normal, signs of sepsis). Most often, an infection of the bladder ascends to the kidneys, causing APN. Symptoms and clinical affection range from mild to severe, but it is always important to recognize and treat APN fast in order to prevent progression to sepsis, renal failure and ultimately death. Uncertain or delayed diagnosis will often lead to an overconsumption of broad-spectrum antibiotics, which contributes to increased development of resistant bacteria and thus threaten the treatment options of the future.

APN diagnosis is primarily made today on the basis of clinical symptoms and findings in the form of flank tenderness, fever and nausea/vomiting. Typical symptoms of cystitis (dysuria, pollakisuria, suprapubic pain, hematuria) are possible but often absent. Especially elderly can present with more generalized signs of infection with nothing clearly indicating localization to the urinary tract. A positive urine culture verifies the diagnosis, but it is only available after a minimum of 24 hours.

To support the diagnosis of an APN and assess its severity, a measure of the systemic inflammatory response is useful such as abnormal temperature, elevated leucocyte count with neutrocytosis, or elevated C-reactive protein (CRP). Some uncertainty is associated with CRP because it has a delayed response to bacterial infection and is often elevated in non-infectious inflammatory conditions. A more sensitive and specific marker is desired that can differentiate between bacterial and viral infection and reflect the severity of the APN. Serum procalcitonin (PCT) has potential as a diagnostic tool in suspected bacterial infections and can distinguish between viral and bacterial urinary infections. Soluble urokinase plasminogen activator receptor (SuPAR) might have a potential as a marker for acute bacterial infections requiring antibiotic treatment. However, there are no well-conducted studies which compare simultaneously all three biomarkers diagnostic abilities for bacterial infections in general or in relation to APN.

The investigators hypothesize that serum CRP, PTC and suPAR have an impact on diagnosing, prognosis, and treatment of patients with a verified APN.

The objectives of the study are:

* To investigate the diagnostic value of CRP, PCT and suPAR in the diagnosis of APN
* To identify the prognostic value of CRP, PCT and suPAR in relation to adverse events in patients with verified APN

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of APN assessed by the receiving physician at the ED

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients with suspected Acute pyelonephritis (APN) from three emergency departments (EDs) in the Region of Southern Denmark (Hospital Sønderjylland, Hospital Lillebælt, Odense University Hospital)
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Verified and non verified acute pyelonephritis (APN) | 2 months after patient discharge
  The decision of whether patients admitted with suspicion of APN actually has a final diagnosis of APN is based on a combination of all findings during admission. The verification of diagnosis requires human handling, interpretation and judgment. Therefore, in this study, an expert panel will define the reference standard for the diagnosis APN. The expert panel consists of two independent consultants from the emergency department with significant experience in emergency medicine and acute infections. They will individually determine whether or not the patient admitted suspected with APN actually had this diagnosis. The final diagnosis will be based on all available relevant information from the patient medical record including MRI of the kidneys. A standardized template will be used. Disagreement will be discussed until a consensus is reached.

SECONDARY OUTCOMES:
Intensive care unit treatment | within 60 days from admission to the emergency department
  transfer to ICU during current admission (binary outcome)
Length of stay | within 60 days from current admission to the emergency department
  days spent in hospital during current admission
The number of participants who died within 30 days | within 30 days from arrival day
  binary - 30-days mortality
The number of participants who died within 90 days | within 90 days from arrival to emergency department
  binary - 90 days mortality
Readmission | within 30 days from day of discharge
  binary
In-hospital mortality | within 60 days from admission to the emergency department
  binary

OTHER OUTCOMES:
Bacteriuria | urine collected within 4 hours of arrival to the emergency department
  Binary outcome defined by microbiologist on urine culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — Hospital of Southern Jutland
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamie L, Daoud G, Nemer G, Nammour T, El Chediak A, Uthman IW, Kibbi AG, Eid A, Kurban M. SuPAR, an emerging biomarker in kidney and inflammatory diseases. Postgrad Med J. 2018 Sep;94(1115):517-524. doi: 10.1136/postgradmedj-2018-135839. Epub 2018 Sep 3. PMID 30177549
- [Background] Schuetz P, Christ-Crain M, Muller B. Procalcitonin and other biomarkers to improve assessment and antibiotic stewardship in infections--hope for hype? Swiss Med Wkly. 2009 Jun 13;139(23-24):318-26. doi: 10.4414/smw.2009.12584. PMID 19529989
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497